CLINICAL TRIAL: NCT06270381
Title: Empower-Grief: Study Protocol for a Pilot Randomized Controlled Trial
Brief Title: Empower-Grief: A Study on a Selective Intervention to Prevent Prolonged Grief Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida (Other)
Responsible Party: Principal Investigator, David#Neto, Principal Investigator, ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UIDB/05299/2020
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Grief Disorder, Prolonged
MeSH Terms: conditions — Prolonged Grief Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants that receive EMPOWER intervention
  Interventions: Other: EMPOWER
- Arm 2 (Active Comparator): Participants that receive treatment as usual (TAU) intervention
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Other: EMPOWER — The EMPOWER intervention (Enhancing and Mobilizing the POtential for Wellness and Emotional Resilience) is a cognitive-behavioral and acceptance-based intervention divided into six modules.In the current application, this intervention is conducted in 6 in-presence or online 50-minute sessions and 2 booster sessions 2 and 4 weeks after the final intervention. It is a manualized treatment in which each session has a specific goal: 1st) Welcome, initial assessment and adherence to the intervention; 2nd) Psychoeducation and transmission of resources for stabilization; 3rd) Psychoeducation on Trauma, Grief and Cognitive-Behavioral Model; 4th)Promoting Experiential Acceptance; 5th) Imagined dialogue; 6th) Coping Training; and two final boosting sessions. In every session, the impact of the previous consultation and evolution is evaluated. This intervention was developed by Lichtenthal et al., 2022.
  Arms: Arm 1
Other: Treatment as usual (TAU) — The treatment as usual (TAU) consists of supportive psychotherapy based on a non-structured and integrative method that focuses on the development of more adaptive coping strategies, understanding and working on the patient's internal models of self, others, and the world. The TAU will be considered during the same period as the EMPOWER intervention.
  Arms: Arm 2

SUMMARY:
The goal of this clinical trial is to test, through a Randomized Controlled Trial (RCT), the efficacy of a selective and short intervention based on second and third-wave cognitive-behavioral interventions (named EMPOWER) for the initial problematic grief reactions and to study potential predictors of adherence and efficacy in bereaved relatives of palliative and oncological patients. The main question is whether EMPOWER intervention is more effective than Treatment as Usual (TAU) in preventing Prolonged Grief Disorder (PGD). Participants with initial indicators of risk of developing PGD will be randomly allocated to EMPOWER and TAU. The primary outcome considered will be symptoms of PGD. The assessment also includes measures of anxiety and depression, attachment, coping, psychological flexibility, posttraumatic growth, and therapeutic alliance. Apart from screening, three assessment moments will be considered: T1: before the first session; T2: at the last session (up to twelve weeks); and T3: follow-up assessment period at 6 months after the previous assessment.

DETAILED DESCRIPTION:
Introduction: Grief reactions of relatives of palliative care patients are seldom addressed. Most interventions focus on Prolonged Grief Disorder (PGD) and not on prevention. This is particularly relevant in palliative and advanced cancer contexts, in which death is the result of a difficult period of a terminal illness making caregivers particularly vulnerable to elevated psychological distress and PGD. Also, matched care interventions align with World Health Organization (WHO)'s (2009) guidelines for organizing mental health services. These guidelines, structured in a pyramid fashion ranging from low-intensity selective interventions and widely available to high-intensity specialized interventions, are tailored to citizens' needs. The differentiation of interventions allows combining need-based timely interventions to prevent PGD while increasing accessibility and mitigating inequality, through rationalization of service delivery.

Aims: The present research intends to implement and evaluate the effectiveness of the low-intensity selective intervention EMPOWER, compared to usual care, in terms of symptoms of prolonged grief and psychological distress in the population of family caregivers who lost a loved one in palliative and advanced cancer contexts. The second objective is to identify predictors of response to intervention. This research is crucial to influence national policy towards a greater emphasis on prevention and early intervention, making the allocation of cost-effective bereavement support services the most efficient and sustainable approach for a significant public health impact in bereavement care.

Procedures: Family members will be contacted from the Centro Hospitalar Universitário Lisboa Norte, by phone, following the usual practice of the clinical service. Those considered at risk, using the cut-off points of risk assessment to be at a moderate level, will be invited to additional intervention and participation in the current study. All participants will provide informed consent before being allocated to one of the two interventions. The informed consent process will cover the study's purpose, procedures, potential risks, and benefits, and it will be obtained from each participant before any data collection or randomization occurs. Participants will be reassured that their data will be anonymized and securely stored. Strategies to enhance participant retention and minimize attrition will be employed, including regular check-ins, reminders for follow-up assessments, a dedicated study coordinator to address participant concerns and flexible scheduling options. Also, a feedback system for participants to express concerns or provide input on the study's procedures will be put in place and this will be used to make necessary adjustments. Throughout their participation, we will emphasize participants' contribution to improving grief support for others and the rigorous privacy and confidentiality measures in place. Treatment will be offered at Centro Hospitalar Universitário Lisboa Norte, local health unit Santa Maria, to family members of patients followed on the palliative care unit and oncology service. To ensure fidelity and quality of intervention delivery across the team the standardized intervention protocol for EMPOWER will be utilized (manualized intervention); providers will receive standardized training and will have ongoing supervision; fidelity assessment tools will be used.

Trial design: a rater-blinded Randomized Controlled Trial (RCT) with two parallel groups, comparing the EMPOWER and treatment as usual (TAU) will take place in order to investigate a two-tier psychological intervention program designed to prevent PGD and offer early intervention for grief-related issues. Randomization will be independently conducted by a research assistant. Participants will be randomly assigned EMPOWER vs. TAU. Randomization will occur after a participant meets eligibility criteria, provides consent, and undergoes risk assessment. The participants will be allocated to each branch of the RCT through block randomization. A random sequence of numbers or allocation codes will be generated using a randomization tool. This sequence will determine the allocation of participants to the two intervention groups. To maintain allocation concealment, the randomization sequence will be securely locked away from researchers involved in recruitment and assessment. When a participant is deemed eligible and has provided informed consent, an independent staff member (or an automated system) not involved in day-to-day study operations will access the randomization sequence to assign the participant. Throughout the study, the project team will continuously monitor the randomization process to ensure it is executed as planned, with any deviations documented and addressed.

ELIGIBILITY:
Inclusion Criteria:

* Having more than 18 years old
* Having experienced the death of a close person (i.e., relative, partner, friend) in the palliative and oncological context
* Having sufficient cognitive abilities and proficiency in the Portuguese language
* Participants will be considered if the death has occurred up to 12 months, considering that the time criterion in diagnosis for prolonged grief disorder is 12 months (and the focus in this study is on prevention)

Exclusion Criteria:

* individuals with a pre-existing severe or active mental disorder predating the loss (e.g., schizophrenia, bipolar disorder, major depression)
* individuals with suicide risk assessed during the intervention
* individuals undergoing other psychological interventions before the loss of the loved one

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Prolonged Grief | pre-first session, last session (up to twelve weeks), follow-up (6 months after the previous assessment)
  Prolonged Grief Scale - Revised (PG13-R). PG13-R is a self-report scale developed by Prigerson et al., (2021) based on DSM-5-TR criteria for PGD. PG-13-R includes 13 items, evaluated in a 5-point likert scale. PG-13-R grief symptoms represent a unidimensional construct, with high degrees of internal consistency in research conducted at Yale (Cronbach's α = .83), Utrecht (Cronbach's α = .90), and Oxford (Cronbach's α = .93) universities. PGD diagnosis is attributed when the person obtains a total value greater than 30 and meets the temporal (12 months) and impairment criteria.

SECONDARY OUTCOMES:
Anxiety and depression | pre-first session; follow-up (6 months after the previous assessment)
  The Hospital Anxiety and Depression Scale (HADS). The HADS measures anxiety and depression symptoms. The scale was developed for non-psychiatric populations (Zigmond & Snaith, 1983). It includes 14 items, evaluated in a 4-point (0-3) likert scale. Values higher than eight in each subscale are suggestive of clinically relevant symptomatology. In a Portuguese sample (Pais-Ribeiro et al., 2007), Cronbach alpha values were .76 in anxiety and .81 in depression.

OTHER OUTCOMES:
Sociodemographic data | screening; pre-first session
  Sociodemographic data include namely age, sex, professional status, education, nationality, marital status, number of children.
Risk Assessment for Grief | screening
  Risk Assessment for Grief (RAG). RAG is a hetero-assessment scale of PGD risk developed by the New Zealand Ministry of Health (Ministry of Health, 2017) and adapted for the DGS norm 003/2019 (DGS, 2019). It includes four items (anger, accusation/guilt, current relationships and general coping with grief) evaluated in a 5-point likert scale. This instrument classifies the degree of PGD risk in low (<7 points), moderate (7-10 points) and high ( ≥ 10 points).
Coping strategies | pre-first session
  BriefCOPE. The BriefCOPE (Carver, 1997) is comprised of 28 items organized into 14 coping strategies. Each coping strategy is measured using two items (humor, positive reframing, emotional social support, acceptance, religion, instrumental support, planning, active coping, behavioral disengagement, self-blaming, substance use, venting, self-distraction; and denial. Participants were asked to answer each item with a Likert-type response scale ranging from 0 (I never do this) to 3 (I always do this). Mean scores were calculated for each coping factor. The study of internal consistency for each factor using Cronbach's alpha shows adequate values (in general α ≤ .60), taking into account there are only two items per factor, for the original (Carver, 1997) and the Portuguese version (Pais Ribeiro & Rodrigues, 2004)
Adult attachment | pre-first session
  Experiences in Close Relationships (ECR-RS). The ECR-RS (Fraley et al., 2011) is self-report instrument that measures adult attachment to relevant persons - in this case the deceased -, rated on a seven-point Likert scale that ranges from 1 (strongly disagree) to 7 (strongly agree). Its 9 items are grouped into 2 dimensions: attachment-related anxiety (items 1-6) and avoidance (items 7-9). The total subscale score consists of the mean of the items and ranges from 1 to 7, with higher scores indicating higher attachment avoidance or anxiety. The Portuguese version showed adequate reliability (α ranged from .72 to .91) and construct validity (Moreira et al., 2015).
Psychological inflexibility | pre-first session
  Acceptance and Action Questionnaire II (AAQ-II). The AAQ (Bond et al., 2011) is a 7-item questionnaire with single-factor structure measuring acceptance, experiential avoidance, and psychological inflexibility. In the Portuguese validation (Pinto-Gouveia et al., 2012) results from a Confirmatory Factor Analysis showed the goodness of fit of the model and this version also demonstrated an excellent level of internal consistency (α=.90) and good convergent and discriminant validity. Individuals are asked to rate each statement on a 7-point Likert scale ranging from 1 (never true) to 7 (always true). This scale reflects the single domain of psychological inflexibility with higher scores indicating greater psychological inflexibility.
Social Support | pre-first session
  The Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS (Zimet et al., 1988) measures perceived social support from family, friends, and others. The 12 items are grouped into 3 factors (family, friends and significant others), each with 4 items, using a 7-point Likert scale (0 = strongly disagree, 7 = strongly agree). Examples of items include "There is a special person who is close by when I need him/her"; "I can talk about my problems with my family". The Portuguese version of the MSPSS (Carvalho et al., 2012) demonstrated good psychometric qualities (α ranged from .85 and .95).
Therapeutic alliance | last session (up to twelve weeks)
  The Working Alliance Inventory-short form (WAI-S). The WAI-S (Tracey & Kokotovic, 1989; Machado & Horvath, 1999 - Portuguese version) is a widely studied 12-item self-report that measures how the client perceives the therapeutic alliance with the therapist, with a 7-point Likert scale ranging from 1 (never) to 7 (always). In addition to the overall alliance score, the WAI-S includes three specific subscales: bond, tasks, and goals (four items, respectively ).
Posttraumatic Growth | follow-up (6 months after the previous assessment)
  Posttraumatic Growth Inventory (PTGI). The PTGI (Tedeschi & Calhoun, 1996) evaluates the extent of perceived positive transformations following a challenging event. Comprising 21 items, it encompasses five subscales: personal strengths, appreciation of life, new possibilities, spiritual changes, and relation to others. Participants were instructed to assess each item on a 6-point Likert scale, ranging from 1 to 6 The overall PTGI score represents the sum of all items and higher scores indicated higher levels of posttraumatic growth. The original version of the PTGI has shown excellent internal reliability (Cronbach's α = 0.90), and acceptable test-retest reliability (r = .71). The PTGI has also shown good psychometric properties in breast cancer Portuguese samples (e.g., Silva et al., 2009).

CONTACTS AND LOCATIONS:
Overall Officials: David Neto, Principal Investigator — ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida
Locations (1):
- Unidade Local de Saúde Santa Maria, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Carvalho, S., Pinto-Gouveia, J., Pimentel, P., Maia, D., & Mota-Pereira, J. (2011). Características psicométricas da versão portuguesa da escala multidimensional de suporte social percebido (multidimensional scale of perceived social support-mspss). Psychologica, 54, 331-357.
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Fraley RC, Heffernan ME, Vicary AM, Brumbaugh CC. The Experiences in Close Relationships-Relationship Structures questionnaire: a method for assessing attachment orientations across relationships. Psychol Assess. 2011 Sep;23(3):615-25. doi: 10.1037/a0022898. PMID 21443364
- [Background] Machado P. P., Horvath A. (1999). Inventário da aliança terapêutica (WAI). In Simões M.R., Gonçalves M. M., Almeida L. S. (Eds.), Testes e provas psicológicas em Portugal (Vol. 2, pp. 87-94). Braga, AP-PORT/SHO.
- [Background] Ministry of Health. 2017. Te Ara Whakapiri: Principles and guidance for the last days of life. (2nd ed). Wellington: Ministry of Health.
- [Background] Moreira H, Martins T, Gouveia MJ, Canavarro MC. Assessing adult attachment across different contexts: validation of the Portuguese version of the experiences in Close Relationships-Relationship Structures questionnaire. J Pers Assess. 2015;97(1):22-30. doi: 10.1080/00223891.2014.950377. Epub 2014 Aug 30. PMID 25175516
- [Background] Pais-Ribeiro J, Silva I, Ferreira T, Martins A, Meneses R, Baltar M. Validation study of a Portuguese version of the Hospital Anxiety and Depression Scale. Psychol Health Med. 2007 Mar;12(2):225-35; quiz 235-7. doi: 10.1080/13548500500524088. English, Portuguese. PMID 17365902
- [Background] Pinto-Gouveia, J., Gregório, S., Dinis, A., & Xavier, A. (2012). Experiential avoidance in clinical and non-clinical samples: AAQ-II Portuguese version. International Journal of Psychology and Psychological Therapy, 12(2), 139-156.
- [Background] Prigerson HG, Boelen PA, Xu J, Smith KV, Maciejewski PK. Validation of the new DSM-5-TR criteria for prolonged grief disorder and the PG-13-Revised (PG-13-R) scale. World Psychiatry. 2021 Feb;20(1):96-106. doi: 10.1002/wps.20823. PMID 33432758
- [Background] Ribeiro, J. L. P., & Rodrigues, A. P. (2004). Questões acerca do coping: A propósito do estudo de adaptação do Brief Cope. Psicologia, Saúde e Doenças, (1), 3-15.
- [Background] Silva, S., Moreira, H., Pinto, S., & Canavarro, M. C. (2009). Cancro da mama e desenvolvimento pessoal e relacional: Estudo das características psicométricas do Inventário de Desenvolvimento Pós-Traumático (Posttraumatic Growth Inventory) numa amostra de mulheres da população portuguesa. Revista Iberoamericana de Diagnóstico e Avaliação Psicológica, 28(2), 105-133.
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Zimet, G. D., Dahlem, N. W., Zimet, S. G., & Farley, G. K. (1988). The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment, 52(1), 30-41. https://doi.org/10.1207/s15327752jpa5201_2
- [Background] Tracey, T. J., & Kokotovic, A. M. (1989). Factor structure of the Working Alliance Inventory. Psychological Assessment: A Journal of Consulting and Clinical Psychology, 1(3), 207-210. https://doi.org/10.1037/1040-3590.1.3.207
- [Background] Lichtenthal WG, Viola M, Rogers M, Roberts KE, Lief L, Cox CE, Brewin CR, Xu JC, Maciejewski PK, Pan CX, Coats T, Ouyang DJ, Rabin S, Vaughan SC, Breitbart W, Marenberg ME, Prigerson HG. Development and preliminary evaluation of EMPOWER for surrogate decision-makers of critically ill patients. Palliat Support Care. 2022 Apr;20(2):167-177. doi: 10.1017/S1478951521000626. PMID 34233779